CLINICAL TRIAL: NCT02503735
Title: Effect of Ledipasvir and Sofosbuvir on Proteinuria and Estimated Glomerular Filtration Rate in Patients With Early Stage (1-3) Hepatitis C Associated Chronic Kidney Disease
Brief Title: Effect of Harvoni on Proteinuria and eGFR in Hepatitis C Virus Associated Chronic Kidney Disease (CKD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment goal
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Raymond Chung, Director of Hepatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-337-1777
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis C; Chronic Kidney Disease
Keywords: CKD; HCV
MeSH Terms: conditions — Hepatitis C; Renal Insufficiency, Chronic | interventions — Sofosbuvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 12 weeks treatment with Sofosbuvir/Ledipasvir (400mg/90mg) (Other): 10 patients with hepatitis C (HCV) and HCV-associated CKD that will receive 12 weeks treatment with Sofosbuvir/Ledipasvir (400mg/90mg)
  Interventions: Drug: Sofosbuvir/Ledipasvir FDC

INTERVENTIONS:
Drug: Sofosbuvir/Ledipasvir FDC — 12 weeks treatment with Harvoni
  Other Names: Harvoni

SUMMARY:
Treatment protocol to see if people with hepatitis C (HCV) and chronic kidney disease (CKD) who are treated with Harvoni for 12 weeks have improvements in their kidney disease.

DETAILED DESCRIPTION:
The investigators hypothesize that patients with early stage (1-3) CKD caused by HCV infection will have significantly improved proteinuria and eGFR after viral eradication with 12 weeks of treatment Harvoni (LDV/SOF). This trial data will serve as the basis to support further study of LDV/SOF in patients with early CKD. Slowing progression of CKD is a critical goal, as the increasing incidence and prevalence of advanced CKD and end stage renal disease (ESRD) places significant health burden on patients and tremendous costs on our health-care system.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed the written informed consent
* Male or female ≥ 18 year of age
* HCV genotype 1 or 4 with ribonucleic acid (HCV RNA) greater than 1000 international units (IU)/milliliter (mL), determined by HCV RNA polymerase chain reaction Roche TaqMan quantitative assay.
* Initial diagnosis of proteinuric chronic kidney disease occurred < 7 years prior to completion of screening
* Women of childbearing potential (i.e. women who have not undergone hysterectomy or bilateral oophorectomy, or no medically documented ovarian failure, and are ≤ 50 years of age) must agree to 1 medically approved contraceptive measures and have their partners agree to an additional barrier method of contraception for the duration of the study and for 4 weeks after the last administration of the study drug. Women of childbearing potential must not rely on hormone-containing contraceptive as a form of birth control during the study but may use. An intrauterine device, female barrier methods with cervical cap or diaphragm with spermicidal agent, tubal sterilization, or vasectomy in male partners.
* Male subjects must agree to consistently and correctly use a condom during heterosexual intercourse and avoid sperm donation for the duration of this study and for 90 days after the last dose of ledipasvir and sofosbuvir. Additionally, if their female partner is of childbearing potential (as defined above), their partner must agree to use either 1 of the non-hormonal methods of birth control listed above or a hormone-containing contraceptive for 90 days after last study drug date. Hormone-containing contraceptive options for partners include implants of levonorgestrel, injectable progesterone, oral contraceptives, contraceptive vaginal ring, or transdermal contraceptive pat
* Adequate organ function defined as follows platelets ≥ 50 x 109/L; hemoglobin ≥ 9 g/dL, estimated glomerular filtration rate ≥ 30mL/min/1.73m2 as estimated by CKD-Epi equation.
* Liver imaging to exclude hepatocellular carcinoma (HCC) is required within 6 months in any patient with cirrhosis.
* Has > 300mg/g creatinine proteinuria on two urine samples obtained within 30 days of starting ledipasvir and sofosbuvir.

Exclusion Criteria:

* History of evidence of clinically significant disorder other than hepatitis C virus infection or clinically significant laboratory finding that in the investigator's judgment would pose a risk to subject safety, interfere with study procedures, or prevent completion of the study.
* Pregnant or lactating female
* Uncontrolled depression or psychiatric disease interfering with the ability to comply with the study procedures or complete the study
* History or presence of any form of cancer within 3 years prior to enrollment, with the exception of excised basal cell or squamous cell carcinoma of the skin, stage 0 or 1 melanoma, or cervical carcinoma in site or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis.
* Experience life-threatening cryoglobulinemic vasculitis requiring initiation of rituximab, steroids or plasmapheresis.
* Concomitant use of cimetidine, trimethoprim or other drugs which can increase tubular creatinine reabsorption
* Uncontrolled cardiovascular or pulmonary disease
* Uncontrolled hypertension
* Known HIV infection
* Known hypersensitivity to ledipasvir or sofosbuvir
* Prior HCV treatment failure using a medication in the NS5A inhibitor class
* Individuals who are taking the following medications and require continuation of the medications during the proposed study period will be excluded, given known interactions with ledipasvir-sofosbuvir: Carbamazepine, phenytoin, phenobarbital, oxcarbazepine, rifabutin, rifampin, isoniazid, rifapentine, rosuvastatin, proton pump inhibitors, digoxin, modafinil, and St. John's wort, milk thistle, Echinacea.
* Having an alternate explanation of chronic kidney disease, including:

  * Diabetic kidney disease, either by biopsy findings or duration of uncontrolled diabetes > 8 years without serologic evidence of immune-complex related kidney disease
  * Chronic hypertensive nephropathy without proteinuria
  * Lupus nephritis
  * Multiple myeloma
  * Obesity related proteinuria, BMI > 35
  * Ongoing nephrotoxic medication use, including NSAIDS
  * Polycystic kidney disease
  * Kidney biopsy showing an alternate explanation for chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hohmann, MD, Study Chair — Chair and Physician Director, Partners Human Research Committees
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Stevens LA, Coresh J, Schmid CH, Feldman HI, Froissart M, Kusek J, Rossert J, Van Lente F, Bruce RD 3rd, Zhang YL, Greene T, Levey AS. Estimating GFR using serum cystatin C alone and in combination with serum creatinine: a pooled analysis of 3,418 individuals with CKD. Am J Kidney Dis. 2008 Mar;51(3):395-406. doi: 10.1053/j.ajkd.2007.11.018. PMID 18295055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 patients were recruited and signed informed consent
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Sofosbuvir/Ledipasvir FDC: 12 weeks treatment with Harvoni (10 total dosed on protocol)
Period: Overall Study
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Started (10/14 consented patients started treatment with Sofosbuvir/Ledipasvir (4 screen failures)) | 10
SVR 12 (12week Post Treatment RNA Neg) | 8
Completed (All 10 subjects who initiated treatment completed treatment) | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Sofosbuvir/Ledipasvir (400mg/90mg) FDC: 12 weeks treatment with Harvoni for patients with Hepatitis C (HCV) and HCV-associated CKD
  Subjects were followed for one year after treatment initiation
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
HCV genotype [Count of Participants; unit: Participants]
  1a | 3
  1b | 4
  4 | 2
  mixed | 1
CKD stage [Count of Participants; unit: Participants]
  1 | 3
  2 | 2
  3 | 5
Baseline HCV RNA [Median (Inter-Quartile Range); unit: IU/mL] | 1,573,500 [564,250 to 4,162,500]
Prior PEG-IFN/ribavirin treatment [Count of Participants; unit: Participants] | 4
Hypertension [Count of Participants; unit: Participants] | 9
Diabetes mellitus [Count of Participants; unit: Participants] | 5
Coronary artery disease [Count of Participants; unit: Participants] | 2
Congestive heart failure [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change in Proteinuria
Description: % change in proteinuria from baseline (timepoint week 0) through timepoint week 24, which was 12 weeks after completion of Harvoni.
Time Frame: Baseline and 24 weeks (12 weeks after completion of Harvoni)
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Participants received sofosbuvir/Ledipasvir FDC for 12 weeks treatment (10 total dosed on protocol)
  Proteinuria is assessed at baseline (initiation of treatment) and at 24 weeks after baseline (12 weeks after completion of treatment.
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 10
percentage change from baseline | -14 [-42 to 52]

2. Secondary Outcome: Median Change in eGFR From Baseline to Timepoint Week 24
Description: Median change from baseline (timepoint week 0) to timepoint week 24, which was 12 weeks after completion of Harvoni.
  Median change in eGFR was calculated using the creatinine and cystatin C-based estimating equation.
  eGFR = 135 × min(SCr/κ, 1)α × max(SCr/κ, 1)-0.601 × min(Scys/0.8, 1)-0.375 × max(Scys/0.8, 1)-0.711 × 0.995Age × 0.969 [if female] × 1.08 [if black]
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m^2
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Participants received sofosbuvir/Ledipasvir FDC for 12 weeks treatment (10 total dosed on protocol)
  We determined the median change in eGFR as measured by creatinine and cystatin C equation from baseline to timepoint week 24 (12 weeks after completion of treatment)
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 10
mL/min/1.73m^2 | 1 [-1 to 2.75]

3. Secondary Outcome: Number of Participants With ≥25% Reduction in Proteinuria
Description: Number of participants with at least -25% change in proteinuria, calculated from baseline (timepoint week 0) to timepoint week 24, which is 12 weeks after completion of Harvoni.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Participants received Sofosbuvir/Ledipasvir FDC for 12 weeks treatment (10 total dosed on protocol)
  We want to determine the number of participants with at least a 25% Reduction in Proteinuria
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 10
Participants | 3

4. Secondary Outcome: Mean Time in Weeks to Maximum Reduction in Proteinuria
Description: This outcome evaluated all post-baseline proteinuria values through the 52 week followup, and determined which demonstrated the greatest negative change (reduction) from baseline. We then calculate the mean time to maximum reduction of proteinuria.
Time Frame: 52 weeks
Population: Because 3 patients had rising proteinuria they are not included in this analysis, which only looks at the mean time to reduction in proteinuria in the 7 patients who had any reductions in proteinuria. This includes the 3 patients who had -25% change in proteinuria and 4 patients who had smaller negative changes (reductions) in proteinuria.
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Participants received sofosbuvir/Ledipasvir FDC for 12 weeks treatment (10 total dosed on protocol)
  The time to maximum reduction in proteinuria was assessed for each participant and compiled, and a mean is presented
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 7
weeks | 39.4 (12.7)

5. Secondary Outcome: Median Change in eGFR From Baseline to Timepoint Week 52
Description: Median change from baseline (timepoint week 0) to timepoint week 52, which was 40 weeks after completion of Harvoni.
  Median change in eGFR was calculated using the creatinine and cystatin C-based estimating equation.
  eGFR = 135 × min(SCr/κ, 1)α × max(SCr/κ, 1)-0.601 × min(Scys/0.8, 1)-0.375 × max(Scys/0.8, 1)-0.711 × 0.995Age × 0.969 [if female] × 1.08 [if black]
Time Frame: 52 weeks
Population: Sofosbuvir/Ledipasvir FDC: 12 weeks treatment with Harvoni (10 total dosed on protocol)
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m^2
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Participants HCV and proteinuria received 12 weeks treatment with Sofosbuvir/Ledipasvir (400mg/90mg)
  The median change in eGFR from baseline to timepoint week 52 was determined, as measured by the creatinine and cystatin C-based estimating equation
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 10
mL/min/1.73m^2 | -4 [-11.25 to 2]

6. Secondary Outcome: Change in Urinary β-2microglobulin Levels Before Therapy
Description: Change in urinary β-2microglobulin levels before therapy with ledipasvir/sofosbuvir fixed dose combination pill.
  β-2microglobulin (mcg/L) change prior to initiating HCV-treatment.
  This outcome was not assessed.
Time Frame: 24 weeks
Population: Data were not collected and the outcome cannot be reported. Values for urinary β-2microglobulin were obtained at baseline and not at screening. Thus we are unable to report a "change in urinary β-2microglobulin levels BEFORE therapy with ledipasvir/sofosbuvir" - however, we are able to report the changes after therapy as followup values were done.
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): 12 weeks treatment with Sofosbuvir/Ledipasvir (400mg/90mg) for patients with HCV and HCV-associated CKD
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Urinary β-2microglobulin Levels After Therapy
Description: Change in urinary β-2microglobulin levels after therapy with ledipasvir/sofosbuvir fixed dose combination pill
  β-2microglobulin (mcg/L) levels were assessed at baseline (timepoint week 0) and at timepoint week 24. Change was recorded for each patient, and presented as a median with IQR.
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: mcg/L
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Participants with HCV and proteinuria received 12 weeks treatment with Sofosbuvir/Ledipasvir (400mg/90mg)
  Change in urinary β-2microglobulin levels after therapy with ledipasvir/sofosbuvir fixed dose combination pill
  β-2microglobulin (mcg/L) levels were measured at baseline and at timepoint week 24
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
Number analyzed (Participants) | 10
mcg/L | 57 [-14 to 546]

ADVERSE EVENTS:
Time Frame: Data was collected over 52 week study period (which includes 12 weeks of treatment with Harvoni, and 40 weeks of post-treatment follow-up).
Groups:
- 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg): Sofosbuvir/Ledipasvir FDC: 12 weeks treatment with Harvoni (10 total dosed on protocol)
  Patients were followed for one year following treatment initiation
Arm/Group | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg) (N=10)
intestinal blockage (Gastrointestinal disorders) | 1 (1) — This severe adverse event (SAE) required hospitalization occurred 4 weeks after completing LDV/SOF. The intestinal condition was pre-existing and the SAE was deemed unrelated to study participation by the principal investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 Weeks Treatment With Sofosbuvir/Ledipasvir (400mg/90mg) (N=10)
fatigue (General disorders) | 3 (4)
nausea (General disorders) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
headache (General disorders) | 2 (2)
reduced appetite (Gastrointestinal disorders) | 1 (1)
acid reflux (Gastrointestinal disorders) | 1 (2)
back/joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
elevated blood prsesure (Vascular disorders) | 1 (1)
mouth pain (Musculoskeletal and connective tissue disorders) | 1 (1)
forgetfulness (Psychiatric disorders) | 1 (1)
frequent urination (Renal and urinary disorders) | 1 (1)
elevated creatinine (Renal and urinary disorders) | 1 (1)
fall / twisted ankle (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT02503735/Prot_000.pdf